CLINICAL TRIAL: NCT02319200
Title: PRIMARY PREVENTION OF HEPATOCELLULAR CARCINOMA BY METFORMIN IN PATIENTS WITH VIRAL C CIRRHOSIS : PROSPECTIVE MULTICENTER STUDY, RANDOMIZED CONTROL TRIAL. Ancillary Study of the ANRS CO12 CirVir Cohort
Brief Title: Primary Prevention Hepatocellular Carcinoma by Metformin
Acronym: METFOVIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision of investigator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P120138
Record Dates: First submitted 2014-12-13; First posted 2014-12-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C, Chronic; Cirrhosis
Keywords: Chemoprevention; Decompensation of cirrhosis; Hepatocellular Carcinoma; Death; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C, Chronic; Fibrosis; Death | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): 1000 mg (2x500 mg) at morning and 1000 mg (2x500 mg) at afternoon (2000 mg per day)
  Metformin daily during 36 months
  Interventions: Drug: Metformin
- placebo tablet (Placebo Comparator): 2 tablets at morning and 2 tablets at afternoon 4 tablets per day
  Interventions: Drug: placebo tablet

INTERVENTIONS:
Drug: Metformin — 1000 mg (2x500 mg) at morning and 1000 mg (2x500 mg) at afternoon (2000 mg per day)
  Metformin daily during 36 months
  Other Names: Glucophage
  Arms: Metformin
Drug: placebo tablet — 4 tablets per day for 36 months
  Arms: placebo tablet

SUMMARY:
Metformin treatment during 36 months could be associated with decreased risk of HCC occurrence and liver related death in patients with compensated HCV cirrhosis and insulinoresistance.

This study is an ancillary of the observational study from the CIRVIR cohort in which more than 1200 patients with compensated HCV cirrhosis are currently included.

participating centers : 26

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is currently the first cause of death of patients with compensated HCV cirrhosis.Despite progresses,existing therapies are limited in their ability to prevent recurrences. Even diagnosed at early stage, long-term prognosis remains poor due to the high rate of recurrence after local treatments. Liver transplantation the only long-term curative treatment is limited by advanced age, comorbidities or the shortage of the graft It concerns less than 5 % of HCC patients . Therefore, the best approach to reduce mortality remains the reduction of HCC incidence.

Abundant observational studies have related a relation between insulinoresistance occurrence and outcome of many cancers. The level of IR assessed by the HOMA index have been recognized as an independent predictive factor of HCC occurrence in patients with compensated viral C cirrhosis. Metformin, a Type 2 diabetic treatment drug, inhibits hepatic gluconeogenesis and increases the stimulation of the glucose uptake in muscle.

Independently of its' anti diabetic effects, Metformin is credited of anti tumoral, anti oxidant, anti inflammatory, and anti angiogenic properties.

Amount epidemiological and experimental data have demonstrated the anti tumoral and chemopreventive effect of metformin in certain cancers.

From our cohort of patients with compensated HCV cirrhosis and not treated by insulin, we have observed that the level of IR assessed by the HOMA was a strong and independent risk factor of HCC occurrence and liver related death. We have also observed in our cohort of diabetic patients with compensated HCV cirrhosis, that treatment by Metformin was associated with a decreased risk of HCC occurrence and liver related death.

HYPOTHESIS

Treatment with metformin could decreased the HCC occurrence and liver related death or transplantation.

MAIN OBJECTIVE

Evaluation the impact of Metformin treatment on HCC occurrence and liver related death in patients with compensated HCV cirrhosis and Insulinoresistance SECONDARY OBJECTIVE

* Occurrence of decompensation of the cirrhosis (ascite, sepsis, encephalopathy, haemorrhage)
* Evaluation of the treatment tolerance

MAIN CRITERION JUDGMENT

Rate of HCC occurrence or liver related-death or transplantation.

SECONDARY CRITERION JUDGMENT

* Occurrence of decompensation of the cirrhosis (ascite, sepsis, encephalopathy, haemorrhage),
* Tolerance

STUDY ASSESSMENTS

The patient of CIRVIR cohort meeting the inclusion criteria will be invited to participate to this study.

During their next visit, the hepatologist, will give full verbal and written information regarding the objective procedures of the study and the possible benefice and side effects of the treatment. A write informed consent will be obtained from all patients who agree to participate to the study.

The treatment period will begin following randomization. On day M0 baseline measurements will be taken and recorded, and metformin administration will be begun. In order to optimize the treatment tolerance, it will be suggested to the patients to take the pill during or at the end of the lunch. During the first week, the posology of the placebo and metformin will be 500 mg at the breakfast. After, the posology will be increased every week as follow: 500 mg morning and afternoon, then 1000 mg morning and afternoon (2000 mg per day). In case of intolerance, the maximum posology tolerated will be maintained. In fact regarding the primary data of the trial regarding the effect of metformin on colonic polyp, it seems possible that low dose of metformin are potentially active This treatment will continue until the end of the study.

FOLLOW UP

Patients will be seen at one month and followed every 3 months. Clinical evaluation and HCC screening are planed In CIRVIR cohort study, Every 6 months.

Duration of Treatment per patient:

• 36 months

Duration of Trial Recruitment:

• 24 months

PARTICIPATING CENTERS : 26

NUMBER OF SUBJECT

In order to demonstrate a reduction of 40% (HR 0.6) of events under metformin vs placebo with 80% power and 5% two-sided alpha risk, 200 patients per arm are necessary.A sample size reassessment will be made after 50% and 75% of patients included based on predictive power calculation.

We estimated that 5% of patients will not tolerate the treatment in the first month, and that 5% more will be lost to follow or not compliant to treatment during the follow up period. Therefore, the number of patients to be included is 222 patients per group.

STATISTICAL ANALYSIS

Clinical data of all the patients will be prospectively collected in a computerized database

Populations analyzed The main analysis will be based on the intent-to-treat population (ITT) of all randomized patients

In addition an explanatory analysis (PP) of all patients randomized & treated without major protocol violations/deviations will be carried out. Pre-defined major protocol violations/deviations are:

1. missing data for the primary efficacy endpoints
2. no study drug received
3. violation of inclusion criteria
4. Additional protocol violations will be possibly defined during the blind data review

Statistical tests. Main criterion: rate of HCC occurrence and liver related-death or transplantation.

The cumulative incidence of HCC and liver-related death or transplantation will be compared according to metformin treatment at inclusion using the log-rank test.

In addition, univariate Cox regression models will be used to identify predictive factors of primary endpoint.

For each endpoint, variables with a P value less than 0.10 in the univariate analysis predicting outcomes will be entered into stepwise Cox regression multivariate models. For sensitivity analyses, the incidence of HCC will be also adjusted on usual risk factors. The same models considering competing risks will be tested using the Fine and Gray test.

Secondary criteria : Occurrence of decompensation of the cirrhosis (ascite, sepsis, encephalopathy, haemorrhage).

Comparisons between groups will be performed first in a univariate manner using the χ2 test or the Fisher-exact tests. Multiple logistic regression models will be used to assessed a possible difference between groups when adjusted on parameters known or identified during the study as possibly affecting these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Patients included in ANRS cohort CO12 CirVir
* Without Hepatic local lesion (s) suggestive of HCC in the inclusion
* No indication for liver transplantation at baseline
* Child Pugh A or B7 at inclusion
* Without co-infection with HIV or HBV
* No history of lactic acidosis or of lactic acidosis at inclusion
* Insulino-resistance: (HOMA ≥2), or Body mass index≥ 25 kg/m ² without diabetes, or untreated known diabetes with HbA1c < 7 %
* No treatment with Metformin or other oral hypoglycemic containing metformin within 30 days before enrollment
* Available healthcare insurance
* Signed written informed consent.

Exclusion Criteria:

* Patient under guardianship or homeless
* Pregnant or breast-feeding women
* Patients with severe disease (excluding HCV liver disease) may threaten short-term life
* Cirrhosis with Child Pugh score> 7
* An alcohol consumption, higher than 40g / day for men and 30g / day for women
* Type 1 diabetes
* Diabetes treated with metformin
* Diabetes not treated with metformin with HbA1c ≥ 7%
* Hypersensitivity / intolerance in biguanides
* Hypersensitivity to the active substance or to any of the excipients.
* Kidney failure defined by creatinine clearance less than 30 ml/ min (MDRD formula)

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
rate of HCC occurrence and liver related-death or transplantation. | at 6 months

SECONDARY OUTCOMES:
occurrence of liver-related complications (Ascites , gastrointestinal bleeding, encephalopathy) | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Roulot, MD, Principal Investigator — Hospital Avicenne
Locations (1):
- Roulot Dominique, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nkontchou G, Cosson E, Aout M, Mahmoudi A, Bourcier V, Charif I, Ganne-Carrie N, Grando-Lemaire V, Vicaut E, Trinchet JC, Beaugrand M. Impact of metformin on the prognosis of cirrhosis induced by viral hepatitis C in diabetic patients. J Clin Endocrinol Metab. 2011 Aug;96(8):2601-8. doi: 10.1210/jc.2010-2415. Epub 2011 Jul 13. PMID 21752887
- [Background] Sangiovanni A, Prati GM, Fasani P, Ronchi G, Romeo R, Manini M, Del Ninno E, Morabito A, Colombo M. The natural history of compensated cirrhosis due to hepatitis C virus: A 17-year cohort study of 214 patients. Hepatology. 2006 Jun;43(6):1303-10. doi: 10.1002/hep.21176. PMID 16729298
- [Background] N'Kontchou G, Mahamoudi A, Aout M, Ganne-Carrie N, Grando V, Coderc E, Vicaut E, Trinchet JC, Sellier N, Beaugrand M, Seror O. Radiofrequency ablation of hepatocellular carcinoma: long-term results and prognostic factors in 235 Western patients with cirrhosis. Hepatology. 2009 Nov;50(5):1475-83. doi: 10.1002/hep.23181. PMID 19731239
- [Background] Perseghin G, Calori G, Lattuada G, Ragogna F, Dugnani E, Garancini MP, Crosignani P, Villa M, Bosi E, Ruotolo G, Piemonti L. Insulin resistance/hyperinsulinemia and cancer mortality: the Cremona study at the 15th year of follow-up. Acta Diabetol. 2012 Dec;49(6):421-8. doi: 10.1007/s00592-011-0361-2. Epub 2012 Jan 4. PMID 22215126
- [Background] Goodwin PJ, Ennis M, Pritchard KI, Trudeau ME, Koo J, Taylor SK, Hood N. Insulin- and obesity-related variables in early-stage breast cancer: correlations and time course of prognostic associations. J Clin Oncol. 2012 Jan 10;30(2):164-71. doi: 10.1200/JCO.2011.36.2723. Epub 2011 Dec 12. PMID 22162568
- [Background] Nkontchou G, Bastard JP, Ziol M, Aout M, Cosson E, Ganne-Carrie N, Grando-Lemaire V, Roulot D, Capeau J, Trinchet JC, Vicaut E, Beaugrand M. Insulin resistance, serum leptin, and adiponectin levels and outcomes of viral hepatitis C cirrhosis. J Hepatol. 2010 Nov;53(5):827-33. doi: 10.1016/j.jhep.2010.04.035. Epub 2010 Jul 14. PMID 20728234
- [Background] Salmon D, Bani-Sadr F, Loko MA, Stitou H, Gervais A, Durant J, Rosenthal E, Quertainmont Y, Barange K, Vittecoq D, Shoai-Tehrani M, Alvarez M, Winnock M, Trinchet JC, Dabis F, Sogni P. Insulin resistance is associated with a higher risk of hepatocellular carcinoma in cirrhotic HIV/HCV-co-infected patients: results from ANRS CO13 HEPAVIH. J Hepatol. 2012 Apr;56(4):862-8. doi: 10.1016/j.jhep.2011.11.009. Epub 2011 Dec 13. PMID 22173166
- [Background] Svegliati-Baroni G, Faraci G, Fabris L, Saccomanno S, Cadamuro M, Pierantonelli I, Trozzi L, Bugianesi E, Guido M, Strazzabosco M, Benedetti A, Marchesini G. Insulin resistance and necroinflammation drives ductular reaction and epithelial-mesenchymal transition in chronic hepatitis C. Gut. 2011 Jan;60(1):108-15. doi: 10.1136/gut.2010.219741. Epub 2010 Oct 21. PMID 20966027